CLINICAL TRIAL: NCT04078360
Title: Alcohol Use Disorders- Mobile Based Brief Intervention Treatment (AMBIT) Technology Innovation to Bridge the Treatment Gap for Hazardous Drinking: A Pilot RCT
Brief Title: Alcohol Use Disorders- Mobile Based Brief Intervention Treatment (AMBIT): A Pilot RCT
Acronym: AMBIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sangath (Other)
Responsible Party: Principal Investigator, Abhijit Nadkarni, Associate Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MR/P020348/1
Record Dates: First submitted 2019-08-28; First posted 2019-09-06 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Hazardous Drinking
Keywords: Hazardous Drinking, mHealth, India, Brief intervention
MeSH Terms: interventions — Ethanol; Methods

STUDY DESIGN:
Intervention Model Description: This will be a parallel three-arm single blind individually randomised controlled trial, with a nested qualitative study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The PI and outcomes assessor will be masked. The screeners will recruit participants into the study, who will then be randomised to one of the three arms of the study. The data team will then assign a masked outcome assessor to collect outcome data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mobile-based intervention (AMBIT) (Experimental): This arm will receive a mobile based program delivered over messages/IVR calls.
  Interventions: Behavioral: AMBIT (Alcohol use disorders- mobile based Brief Intervention treatment) intervention
- Face-to-face counselling (Active Comparator): This arm will receive a brief counselling session from a trained health worker.
  Interventions: Behavioral: Face to face Brief Intervention
- Active control (Active Comparator): This arm will receive an educational BI leaflet.
  Interventions: Behavioral: BI leaflet intervention

INTERVENTIONS:
Behavioral: AMBIT (Alcohol use disorders- mobile based Brief Intervention treatment) intervention — The intervention will consist of participants receiving messages and/IVR calls not more than twice or thrice a week on their mobile phone for a duration of 8 weeks. Messages/IVR calls will be sent through VIAMO's technology platform. Each week messages will be focussed on specific content areas derived from the formative research of the study. Some of the components of the intervention include:
  1. Self awareness messages
  2. Self reflection messages
  3. Motivational messages
  4. Messages on safe drinking, alcohol reduction, drinking management, risk management, craving management and drinking alternatives.
  5. Health education messages
  6. Personalized feedback and information
  7. Help-seeking resources
  8. Goal setting messages
  Arms: Mobile-based intervention (AMBIT)
Behavioral: Face to face Brief Intervention — The intervention will consist of the participants receiving the BI based on the WHO Mental Health Gap Action Programme (mhGAP) intervention from a trained researcher. The BI will be conducted over a single session (5-10 mins).
  Arms: Face-to-face counselling
Behavioral: BI leaflet intervention — The intervention will consist of an educational BI leaflet consisting of health information on alcohol consumption, and tips to manage and reduce drinking.
  Arms: Active control

SUMMARY:
The World Health Organization (WHO) defines three levels of problematic alcohol use; hazardous drinking (HD) (which puts a person at risk of developing health/social problems), harmful drinking (where health/social problems are already occurring), and alcohol dependence (where serious problems have already occurred). Although HD and harmful drinking affects a larger proportion of the population (and causes many more problems) than alcohol dependence, Indian health policy focuses mainly on institutional delivery of care for alcohol dependence. Extensive evidence globally demonstrates the effectiveness of Brief Interventions (BIs) in reducing drinking in HD. However, in India, barriers to providing such treatments are the inequitable distribution of trained healthcare professionals and concerns about the cultural generalisability of interventions developed in the West. Mobile phone technology like SMS (Short Messaging Service) and interactive voice response (IVR) can deliver BIs to large numbers of HDs, quickly and at low cost, as demonstrated in smoking cessation interventions. Furthermore, a growing body of evidence demonstrates that following a systematic methodology to culturally adapt psychosocial interventions increases acceptability by recipients and delivery agents, and feasibility of delivery. The overall objective of AMBIT is to develop a contextually appropriate BI for HD that can be delivered using mobile phone technology to overcome barriers to access in low resource settings.

Preliminary formative research has informed the development of the first version of the treatment package, which was tested through a case series, by refining the intervention content and delivery through an iterative process, to develop the final intervention. This pilot Randomised Control Trial (RCT) will aim to empirically evaluate the feasibility and acceptability, as well as preliminary impact of the BI, and fine-tune the procedures for a definitive RCT. It therefore does not have clear hypotheses, but instead different primary objectives, which are listed in the following.

OBJECTIVES

1. To assess the feasibility of delivering the mobile-based BI.
2. To assess the acceptability of delivering the mobile-based BI.
3. To inform sample size calculation (based on preliminary estimate of effectiveness) and refine procedures for a definitive RCT.
4. To refine the mobile-based BI package for a definitive RCT.
5. To assess the impact of the mobile-based BI, on treatment outcomes.

DETAILED DESCRIPTION:
The AMBIT study is aimed at developing and evaluating a mobile based BI for hazardous drinkers in Goa-India. The first version of the treatment package was developed through formative research, and tested through a case series, to develop the final intervention. This pilot Randomised Control Trial (RCT) will aim to empirically evaluate the feasibility, acceptability and preliminary impact of the BI, and fine-tune the procedures for a definitive RCT. This protocol will serve as a research framework for the implementation of the proposed pilot RCT.

OBJECTIVES

1. To assess the feasibility of delivering the mobile-based BI.
2. To assess the acceptability of delivering the mobile-based BI.
3. To inform sample size calculation (based on preliminary estimate of effectiveness) and refine procedures for a definitive RCT.
4. To refine the mobile-based BI package for a definitive RCT.
5. To assess the impact of the mobile-based BI, on treatment outcomes. METHODS Study sample- A sample of 120 participants will be recruited; approximately evenly spread out across all study settings and interventions. The sample size is not based on formal power calculations as the study is not designed to test a hypothesis. The sample size estimations have been made based on our previous experiences of pilot RCTs and deemed sufficient to achieve the goals of understanding the acceptability, feasibility, and preliminary impact of an intervention.

Recruitment Procedure- In all three settings, researchers, who will identify hazardous drinkers through appropriate screening procedures. Eligible participants will be invited to join the study if they provide voluntary consent to participate.

In educational institutions and workplaces: At educational institutions and workplaces participant recruitment will be nested within the health and wellness camp (previously tested during the formative research phase), that includes screening for two other health-related issues (Perceived Stress and Physical Activity) aside from AUD screening. This is done to overcome resistance to entering screening for an alcohol-related program, due to cultural stigma around alcohol consumption. It is expected that by introducing screening for a range of health issues, this issue will be mitigated.

In PHCs: The researchers will perform universal screening.

Recruitment will also be done through referrals from the following sources:

* Self: Potential participants will learn about our program through advertising (e.g. banners, posters and leaflets) and then approach a researcher for screening.
* Gatekeepers: (e.g. At Colleges: Faculty/Students; At workplaces: Human Resource [HR] officials/peers; At PHC's: Medical officers and PHC staff): The researchers will seek assistance from these gatekeepers to build awareness about the project, and refer potential participants to the researchers.

Screening tools: All participants will be screened using the AUDIT to identify hazardous drinking (Saunders, 1993). Other tools that will be used as part of the 'Health and Wellness Camp' will include the International Physical Activity Questionnaire (IPAQ) (Booth, 2000), and Perceived Stress Scale (PSS) (Cohen, Kamarck, & Mermelstein, 1983).

AUDIT is a 10 item screening tool developed by the World Health Organisation (WHO) for the detection of AUD. It has been validated in India (Pal et al., 2004), used in cross-national studies, and used in the study setting (Nadkarni, 2017). For a previous study, the AUDIT has been translated into Konkani (Goan vernacular), using a systematic translation-back translation method with two teams of translators, followed by an item-by item analysis and selection by consensus (Silva et al., 2003). The AUDIT is used to identify AUDs and categorise it into hazardous drinking (score of 8-15), harmful drinking (16-19) and dependent drinking (>20) The Perceived Stress Scale (PSS) is a widely used instrument for measuring perception of stress. It has been empirically validated (Lee et al, 2012) with college students and workers and translated into 25 languages.

The International Physical Activity Questionnaire (IPAQ) is widely used to measure health related physical activity, and has acceptable measurement properties for use in many settings and in different languages, and is suitable for use among young and middle-aged adults (15-69 years).(Lee et al, 2011)

Consenting procedures:

All eligible participants will be informed about the study, taken through the informed consent process and requested to provide written consent to participate. The researcher will ensure that any queries about the intervention are resolved. All consent procedures will be audio-recorded with the permission of the participant.

Sampling Procedure- Stratified randomisation will be used. Consenting eligible participants will be stratified into three strata, based on the recruitment site- educational institutions, workplaces and PHCs. Consenting participants from each stratum will be randomized to receive our intervention (AMBIT), face-to-face BI or active control. An independent data manager will generate a randomisation list and participants will be randomised using Sequentially Numbered Opaque Sealed Envelopes to maximise allocation concealment.

Baseline assessments

Baseline measures administered to consenting participants include:

1. Data about potential confounders through a socio-demographic form, such as age, gender, employment status, educational status, and marital status. In addition, we will collect information required for the delivery of the intervention such as preferred days/time to receive the SMS/IVR, preference for SMS and/or IVR (For the participants receiving the mobile-based intervention)
2. TLFB (Time Line Follow Back method): The TLFB is a calendar method of collecting data about quantity and frequency of drinking. The TLFB has high test-retest reliability and concurrent validity has been established in various types of AUD. The TLFB has been used in previous research at the study site (Nadkarni, 2017).

Outcome Assessment:

Adding to the primary and secondary outcomes mentioned in other parts of this registration, process indicators will be collected. These include the following:

* Number of participants screened for AUDs in each setting
* Number and proportion of participants screened positive for HD on AUDIT
* Number and proportion of participants consenting for the treatment
* Number and proportion of dropouts during the 8 week treatment (Dropouts are defined as participants choosing to stop receiving the intervention messages)
* Reasons for refusal to participate
* Reasons for drop-out
* Proportion of participants choosing SMS vs IVR vs both
* Proportion of participants that listen to the complete IVR
* Proportion of participants with high engagement (defined as response to more than 50% of messages).
* Number and proportion of participants completing outcome assessment Nested qualitative study- Qualitative outcome interviews will also be conducted with a sub-sample of participants after outcome assessment to gain insight into the impact of the mobile-based BI on the hazardous drinker. We will purposively select treatment completers and drop-outs, those who reduce drinking and those who do not, to understand their perceptions of the treatment and suggestions to improve the intervention. An interview guide will be developed which focuses on understanding acceptability, feasibility and perceived impact of the mobile based BI.

Monitoring and follow up:

Study researchers will submit a daily log on the challenges faced in recruitment at each site to the project coordinator during recruitment. Researchers will also send information on the number of participants recruited each day to the project data manager as per the daily case reporting form. The coordinator will provide daily supervision via phone call, review the daily logs and visit each site weekly. Any challenges will be addressed by the Project Coordinator over the course of the study.

As soon as a participant is recruited to the mobile-based BI, contact information (excluding name) along with relevant details such as treatment preferences will be shared with VIAMO's project manager. The project data manager will be responsible to upload participant details on VIAMO's platform within 24 hours post-recruitment. Upon receiving study participant details through the VIAMO platform, VIAMO's project manager will be responsible to initiate mobile based intervention with participants no later than 48 hours upon receiving participant details. Accordingly, every participant will receive the mobile based BI for 8 weeks. The data manager and program coordinator will monitor the delivery of the intervention for each participant and export data from the VIAMO platform on a weekly basis.

Data transfer and storage:

oBaseline and outcome data will be collected by the Researcher using the tablet devices which will have pre-programmed check rules. The treatment data will be exported via the VIAMO platform as an excel file on a weekly basis.

oAll data from the VIAMO platform and tablet data will be downloaded weekly on a dedicated computer with internet connection and updated antivirus software.

oCSV data files will be downloaded by site and merged using a CSV file merge utility.

oThe merged file will be saved in a folder (categorised by the week) and backed up on to the server. The weekly file will be additionally backed up on an external hard drive as an additional safety measure.

oThe Data Manager will be responsible for counting and checking the forms received from the sites.

oA log of missing forms or incomplete data (if any) will be reported to the concerned researcher by the Data Manager and the same will be received within two working days.

oVerified paper forms will be entered into STAR software system running on desktops or on an excel spreadsheet.

oAll CSV files will be converted into Excel/SPSS/Stata file format.

Data Storage:

Participant details and confidential information collected on the consent form will be safely stored in a cupboard, which will be locked and the keys will be in the custody of the Data Manager. Secure transfer of the forms from the data team to outcome evaluations team will be done by the data entry assistant.

Data analysis:

Quantitative- Baseline characteristics of individuals who consented and did not consent, and participants who did and did not complete outcome assessments, as will baseline characteristics of participants in the intervention arms versus those in the control arm, will be presented as proportions or means. The process indicators will be presented consistent with CONSORT guidelines (Moher et al, 2001) including a trial flow chart. The primary analysis will be intention-to-treat at the 2 month end-point regardless of treatment adherence, adjusted for baseline AUDIT. Regression analysis will be conducted for the treatment outcomes. Effect sizes will be reported as mean differences and standardised mean differences with 95% confidence intervals for continuous outcomes.

Qualitative- Thematic analysis will be used to analyse the qualitative data from the outcome interviews, using Nvivo version 11. Analysis will involve generation of codes from raw data. Themes will be derived by retrieving pieces of data pertaining to codes and by examining their meaning in relation to the research questions (acceptability of the content and delivery of the mobile-based BI, engagement barriers, impact on drinking).

OUTPUT At the end of the pilot RCT, data obtained will be used to frame a contextually adapted BI for HD that can be further tested for cost effectiveness in a definitive RCT. The learnings from the pilot RCT will be synthesised to refine procedures for a definitive RCT and the preliminary understanding of effect sizes will be used to plan sample size for a subsequent definitive RCT.

ELIGIBILITY:
Inclusion criteria:

* Hazardous drinkers (Alcohol Use Disorder Identification Test [AUDIT] score = 8-15). AUDIT is a 10-item screening questionnaire developed by the WHO for the detection of alcohol use disorders (Saunders et al., 1993).
* Adult (>18 years) males and females in educational institutions
* Males aged 18-65 years in workplaces and primary health centres
* Personal ownership of a mobile phone and is SMS/IVR call savvy.

Exclusion criteria:

* Females (In workplaces and primary health centers)
* Participants owning a shared/family phone
* Aged <18 years and >65 years
* Owns a mobile phone but is not SMS/IVR call savvy
* Harmful and dependent drinkers (AUDIT score >15)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Males are included in all settings (educational institutions, workplaces and primary health centers) Females are included in colleges
Enrollment: 74 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Change in Time Line Follow Back (TLFB) measure of frequency of drinking- Percent Days Abstinent (PDA). | At baseline and at 3 months post-randomisation in all participants regardless of treatment engagement
  TLFB (Time Line Follow Back method): The TLFB is a calendar method of collecting data about quantity and frequency of drinking and various memory aids are used to enhance recall (e.g. special dates).. The TLFB has high test-retest reliability and concurrent validity has been established in various types of AUD. The TLFB has been used in previous research at the study site (Nadkarni, 2017) Percent Days Abstinent reflects on which percentage of 14 days prior to assessment a participant has not drunk any alcohol.

SECONDARY OUTCOMES:
Change in Time Line Follow Back measure of quantity of drinking- gms ethanol/week. | At baseline and at 3 months post-randomisation in all participants regardless of treatment engagement
  Gms ethanol/week: Amount of ethanol consumed per week as measured via Time Line Follow Back method.
Change in Time Line Follow Back measure of patterns of drinking-Percent Days Heavy Drinking (PDHD). | At baseline and at 3 months post-randomisation in all participants regardless of treatment engagement
  Percent Days Heavy Drinking: The percentage of days measured via TLFB on which the participant drank heavily (defined as at least 6 drinks per day).
Change in Time Line Follow Back measure of intensity of drinking-gms ethanol per drinking day. | At baseline and at 3 months post-randomisation in all participants regardless of treatment engagement
  Intensity of drinking - gms ethanol per drinking day: The average amount of ethanol consumed by a participant on drinking days over the 14 days timeframe measured via the TLFB.

CONTACTS AND LOCATIONS:
Overall Officials: Abhijit Nadkarni, MBBS, Principal Investigator — Sangath
Locations (1):
- Goa Police, Panjim, Goa, India

IPD SHARING:
Plan to Share IPD: No